CLINICAL TRIAL: NCT03002285
Title: Evaluation of Speed-accuracy Trade-off in a Computer Task in Individuals With Cerebral Palsy
Brief Title: Fitts Law in People With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14652713.9.0000.0082
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cerebral Palsy group (Experimental): Group with Cerebral Palsy that performed the Fitts law in a computer task
  Interventions: Behavioral: Cerebral Palsy group
- Control group (Active Comparator): Group with typical development that performed the Fitts law in a computer task
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Cerebral Palsy group — Group with Cerebral Palsy that performed the Fitts law in a computer task
  Arms: Cerebral Palsy group
Behavioral: Control group — Group with typical development that performed the Fitts law in a computer task
  Arms: Control group

SUMMARY:
Introduction: Cerebral palsy (CP) is a non-progressive disorder in the brain which makes the control and execution of movements difficult. One of the possible ways to analyze motor control in these individuals could be through analysis of movement speed and accuracy. Objective: To verify the speed-accuracy trade-off in individuals with CP. Method: 96 individuals were evaluated, 48 with CP and 48 with typical development (TD), matched by age and sex. The software used was the "Fitts' Reciprocal Aiming Task v.1.0 (Horizontal)", performed on a computer using an external optical mouse, with progressive indices of difficulty (IDs): ID2, ID4a and ID4b. Each index of difficulty was performed three times and the total time/touches captured.

DETAILED DESCRIPTION:
The software used in this study was "Fitts' Reciprocal Aiming Task v.1.0 (Horizontal)" developed by Okazaki, in the public domain and available on the Internet, which was performed on a Toshiba notebook®, model Satellite A60-S1561 System Unit, with the use of an external optical mouse, Fortrek® OM-302.

This instrument can be used to verify motor control through analysis of the speed and accuracy of movement, which can be determined through the log-linear relation between movement time and task difficulty using a mathematical equation, and analyzed by Fitts' law, which describes the relation between movement accuracy and speed, associated with target size and distance11. Thus, the task used in this study was composed of targets of different sizes, being that the smaller targets require more time to execute due to the necessity of increased accuracy and, if the distance between targets reduces, the speed of movement becomes greater and the accuracy decreases.

In relation to target size (W) and distance between targets (D), the equation log2 (2D/W) results in an index of difficulty (ID), where the higher the ID, the more difficult the task, a fact that necessitates greater movement time.

To evaluate the speed and accuracy, two different indices of difficulty were used in this study (ID2 and ID4). The difficulty level was increased by changing the width and distance between the bars. In addition, ID4 was used in two different ways (ID4a and ID4b), for which the distance between the bars and the width were different, but the ID was maintained.

3 Procedure and design The experiment was composed of three trials at each of the two IDs: 2 and 4 (ID 4 had two kinds of measurement - ID4a and ID4b), and the participants performed the tasks individually in a room, with only the evaluator present, seated on a chair (or their own wheelchair), which was adjusted in height according to the needs of the individual. A footrest was available, when necessary. The computer was placed on a table, and each participant was given instructions and presented with the task, in which the individual, after hearing an alarm from the computer, was required to click with an external mouse cursor on two parallel bars which were arranged vertically, intermittently, with the greatest speed and accuracy possible, for a period of 10 seconds, followed by a second alarm which indicated the end of the attempt.

Directly following the attempt, the total movement time was registered, by dividing the seconds obtained in each attempt by the number of "clicks" on targets. If more than two clicks were wrong, the individual repeated the task.

Procedure and design The experiment was composed of three trials at each of the two IDs: 2 and 4 (ID 4 had two kinds of measurement - ID4a and ID4b), and the participants performed the tasks individually in a room, with only the evaluator present, seated on a chair (or their own wheelchair), which was adjusted in height according to the needs of the individual. A footrest was available, when necessary. The computer was placed on a table, and each participant was given instructions and presented with the task, in which the individual, after hearing an alarm from the computer, was required to click with an external mouse cursor on two parallel bars which were arranged vertically, intermittently, with the greatest speed and accuracy possible, for a period of 10 seconds, followed by a second alarm which indicated the end of the attempt.

Directly following the attempt, the total movement time was registered, by dividing the seconds obtained in each attempt by the number of "clicks" on targets. If more than two clicks were wrong, the individual repeated the task.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of CP;
* levels I to IV according to the GMFCS;
* levels I to III according to MACS.

Exclusion Criteria:

* presence of surgery or a chemical neuromuscular blockade in the upper limbs within six months prior to participation in the study;
* lack of comprehension of the experimental instructions.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Motor control test by using a fitts law task in computational task | one day

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fernani DCGL, Prado MTA, da Silva TD, Massetti T, de Abreu LC, Magalhaes FH, Dawes H, de Mello Monteiro CB. Evaluation of speed-accuracy trade-off in a computer task in individuals with cerebral palsy: a cross-sectional study. BMC Neurol. 2017 Jul 27;17(1):143. doi: 10.1186/s12883-017-0920-4. PMID 28750603